CLINICAL TRIAL: NCT01468597
Title: Does Platelet Inhibition Predict Surgery Related Bleeding in Patients Undergoing Emergent Cardiac Surgery During Dual Antiplatelet Therapy - a Pilot Study
Brief Title: Platelet Inhibition and Bleeding in Patients Undergoing Emergent Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: 21-202 ex 09/10
Record Dates: First submitted 2011-10-04; First posted 2011-11-09 (Estimated); Results first posted 2020-06-18 (Actual); Last update posted 2020-06-18 (Actual); Status verified 2020-06

CONDITIONS: Bleeding
Keywords: Emergent; Cardiac surgery; On-pump; Platelet function
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- One group: Emergency surgery

SUMMARY:
The aim of the study is to evaluate if there is an association between platelet inhibition and surgery-related bleeding in patients undergoing emergent cardiac surgery during dual antiplatelet therapy.

DETAILED DESCRIPTION:
Blood for measuring platelet function is drawn before induction of anesthesia

ELIGIBILITY:
Inclusion Criteria:

* First time on-pump CABG with or without valve replacement

Exclusion Criteria:

* Redo surgery,
* Renal insufficiency needing dialysis,
* Concomitant medication with warfarin,
* Preoperative fibrinogen < 150 mg%

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients needing emergent cardiac surgery under dual antiplatelet therapy
Sampling Method: Non-Probability Sample
Enrollment: 167 (Actual)
Dates: Start 2011-01; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Mahla, M.D., Principal Investigator — Department of Anesthesia and Intensive Care Medicine, Medical University of Graz
Locations (1):
- Department of Anesthesiology and Intensive Care Medicine, Department of Surgery, Medical University of Graz, Graz, Austria

REFERENCES:
- [Derived] Mahla E, Prueller F, Farzi S, Pregartner G, Raggam RB, Beran E, Toller W, Berghold A, Tantry US, Gurbel PA. Does Platelet Reactivity Predict Bleeding in Patients Needing Urgent Coronary Artery Bypass Grafting During Dual Antiplatelet Therapy? Ann Thorac Surg. 2016 Dec;102(6):2010-2017. doi: 10.1016/j.athoracsur.2016.05.003. Epub 2016 Jul 1. PMID 27378554

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 184 patients were screened for eligibility. Of these, 17 patients were found to be ineligible for the study.
  Therefore the number of actually enrolled patients is 167.
Period: Overall Study
Arm/Group | One Group
Started | 184
Completed | 149
Not Completed | 35
Not completed — Found ineligible | 17
Not completed — concomitant valves | 12
Not completed — off-pump CABG | 1
Not completed — no platelet function data | 5

BASELINE CHARACTERISTICS:
Arm/Group | One Group
Number analyzed (Participants) | 149
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.2 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 114
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 149
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Austria | 149

OUTCOME MEASURES:

1. Primary Outcome: Calculated Blood Loss
Time Frame: until postoperative day 5
Measure: Median (Inter-Quartile Range); unit: milliters
Arm/Group | One Group
Number analyzed (Participants) | 149
milliters | 1996 [937 to 1572]

2. Secondary Outcome: BARC Bleeding
Description: Intracranial bleed within 48 hours, Reoperation after closure of sternotomy for the purpose of controlling bleeding, Transfusion of equal to or more than 5 Units of packed red blood cells within a 48-hour period, Chest tube output of equal to or more than 2 L within a 24-h period.
Time Frame: until postoperative day 2
Measure: Number; unit: participants
Arm/Group | One Group
Number analyzed (Participants) | 149
participants | 72

ADVERSE EVENTS:
Arm/Group | One Group
All-Cause Mortality (participants affected / at risk) | 13/149
Serious Adverse Events (participants affected / at risk) | 13/149
Other Adverse Events (participants affected / at risk) | 0/149
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | One Group (N=149)
Mortality (General disorders) | 13 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes